CLINICAL TRIAL: NCT04465383
Title: A Prospective Randomized Controlled Monocentric Study Comparing Digital Sedation Versus Intravenous Sedation Among Patients Undergoing Colonoscopy
Brief Title: Digital Sedation: Virtual Reality Hypnosis During Colonoscopy
Acronym: COLDiS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too complicated during pandemics. Phase 2 of recruitment completed and enough data available.
Sponsor: Oncomfort (Industry)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OC08
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Sedation (Experimental): Digital Sedation with rescue intravenous sedation (propofol) if needed upon patient request
  Interventions: Device: Aqua© 30 on Oncomfort SedakitTM; Drug: Propofol
- Intravenous sedation (Active Comparator): Control arm with conventional Intravenous sedation
  Interventions: Drug: Propofol

INTERVENTIONS:
Device: Aqua© 30 on Oncomfort SedakitTM — Digital Sedation session consists in a virtual reality software (Aqua© 30 Version 3.0, Oncomfort SA, Waver, Belgium) including a clinical hypnosis script.Patients in the intervention group will undergo a 30-minute Digital Sedation program through a VR headset and headphones. This medical device called Oncomfort SedakitTM has been created to reduce anxiety and pain during medical/ surgical interventions
  Arms: Digital Sedation
Drug: Propofol — Standard sedation starting doses of 1 µg/ml to 6 µg/ml depending on patient's reaction and titrated incrementally by 0.5µg/ml. Doses are adapted according to the level of comfort and needs of the patient.

SUMMARY:
This prospective Randomized Controlled Trial will evaluate efficacy, safety, and pharmacoeconomic outcomes in patients undergoing colonoscopy with either Digital Sedation using the Aqua© module of the Oncomfort device (Sedakit TM) or the standard of care, intravenous sedation with propofol. The Aqua© module is designed for sedation and management of pain and anxiety related to medical and surgical procedures.

DETAILED DESCRIPTION:
This prospective Randomized Controlled Trial will evaluate efficacy, safety, and pharmacoeconomic outcomes in patients undergoing colonoscopy with either Digital Sedation using the Aqua© module of the Oncomfort device (Sedakit TM) or the standard of care, intravenous sedation with propofol. The Aqua© module is designed for sedation and management of pain and anxiety related to medical and surgical procedures.

Participants will be recruited during the anesthesiology consultation conducted in preparation for colonoscopy. Those with indication for screening or diagnostic colonoscopy under conventional intravenous sedation (propofol) and willing to participate will provide their written informed consent and will be randomized (2:1) between two arms:

1. Experimental arm: Digital Sedation, with rescue intravenous sedation (propofol) if needed upon patient request
2. Control arm: conventional intravenous sedation (propofol)

The study will be divided into three stages, with randomization (2:1) maintained throughout. In the first stage, accrual will be halted when about 45 patients have been randomized, at least 27 of whom being evaluable patients randomized to the experimental arm. A non-binding futility analysis is planned for the primary outcome. In the second stage, accrual will be halted when about 90 patients have been randomized. A non-binding futility analysis is planned for the primary outcome. If the milestones are met, accrual will be reopened to the second stage and the study will continue to the planned final accrual of 177 patients (118 to experimental and 59 to control arm, respectively). At the end of the recruitment of Stage 1 and 2, an analysis of the secondary outcomes will also be run. Results of these analysis could also impact the decision for pursuing to second/ third stage.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Indication for screening or diagnostic colonoscopy under conventional IVS (propofol)
* Provision of written informed consent

Exclusion Criteria:

* Scheduled dilation
* Active Crohn Disease
* Low auditory acuity that precludes use of the device
* Low visual acuity that precludes use of the device
* Head or face wounds precluding use of the device
* Schizophrenia
* Dizziness
* Water/sea phobia
* Non-proficiency in French or Dutch (research language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
To confirm the feasibility of using digital sedation in colonoscopy (stage 1) | Day 1
  cecal intubation rate, rate of rescue sedation
To demonstrate adequate performance of colonoscopy using digital sedation (stage 2) | Day 1
  cecal intubation rate, rate of rescue sedation

SECONDARY OUTCOMES:
To compare patient experience in both arms | Day 1 & Day 2 Follow-up call
  Measure of satisfaction by Likert scale (0 to 5), pain by Visual Analogue Scale (VAS 0 to 10), anxiety by Visual Analogue Scale (VAS 0 to 10), comfort by Visual Analogue Scale (VAS 0 to 10), Preferred type of sedation, Recall of the procedure, Experienced side effects/ AE
To compare measures of colonoscopy performance in both arms | Day 1
  Compare Cecal intubation rates, Adenoma detection rates, Withdrawal time,Total duration of colonoscopy, Total duration of sedation,Total length of stay in procedure room,Total length of stay in recovery room,Total length of stay in hospital
To assess the need for rescue sedation in the experimental arm | Day 1
  Proportion of patients with cecal intubation without rescue sedation in the experimental arm, Frequency of use of intravenous sedation (propofol) and of complete interruption of digital sedation
To compare use of sedation medication in both arms | Day 1
  Average (per patient) total doses of sedation medication per arm
To assess gastroenterologist and anesthesiologist satisfaction in both arms | Day 1
  Measure of satisfaction by Likert scale (0 to 5) and of perceived facilitation or impediment of the procedure by Digital Sedation as measured by Likert scale (0 to 5)
To assess gastroenterologist and anesthesiologist stress in both arms | Day 1
  Measure of stress by Visual Analogue Scale (VAS 0 to 10)
To compare physiologic measures in both arms | Day 1
  Oxygen saturation (minimal observed during procedure), MBP (min/max.), Heart rate (min/max)
To assess difficulty or ease of the procedure in both arms | Day 1
  Number of abdominal manipulations and patient mobilizations
To compare the safety in both arms | Screening, Day 1 & Day 2 Follow-up call
  Frequency and type of AEs and SAEs, Frequency and severity of episodes of desaturation and of HR/ MBP changes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blero, Prof. MD., Principal Investigator — Erasme University Hospital
Locations (1):
- Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No